CLINICAL TRIAL: NCT04042051
Title: Phase Ib Clinical Trial of Copanlisib in Combination With Trastuzumab Emtansine (T-DM1) in Pretreated Unresectable Locally Advanced or Metastatic HER2-positive Breast Cancer "Panthera"
Brief Title: Copanlisib in Combination With T-DM1 in Pretreated Unresectable Locally Advanced or Metastatic HER2-positive Breast Cancer
Acronym: Panthera
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual rate to date was too low to finish the trial in a reasonable timeframe
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE 17-13
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer; Metastatic Breast Cancer; Locally Advanced Breast Cancer; Unresectable Breast Cancer
Keywords: HER2; HER2-positive; Metastatic; Breast; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — copanlisib; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): This study is a phase Ib open label, single arm, adaptive multi-centre trial. Patients with unresectable locally advanced or metastatic HER2-positive breast cancer who previously received trastuzumab and a taxane, separately or in combination, will be treated with copanlisib (as assigned at registration according to the dose escalation scheme) plus trastuzumab emtansine 3.6mg/kg IV on day 1 of a 21-day cycle.
  Interventions: Drug: Copanlisib; Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Copanlisib — Copanlisib is supplied as lyophilized preparation in a 6mL injection vial. The total amount of copanlisib per vial is 60mg. The solution for IV infusions is obtained after reconstitution with normal saline solution. Copanlisib will be administered on Days 1 (and 8 and 15 [according to the dose escalation scheme]) of each 21-day cycle. Copanlisib will be administered first over 60 minutes followed by the infusion of trastuzumab emtansine.
  Other Names: BAY 80-6946
Drug: Trastuzumab emtansine — Trastuzumab emtansine 3.6mg/kg IV infusion on Day 1 of each 21-day treatment cycle.
  Other Names: Kadcyla

SUMMARY:
This study is a Phase 1b open label, single arm, adaptive multi-centre trial of copanlisib in combination with trastuzumab emtansine (T-DM1) in pretreated locally advanced or metastatic HER2-positive breast cancer.

Patients with unresectable locally advanced or metastatic HER2-positive breast cancer who previously received trastuzumab and a taxane, separately or in combination, will be treated with copanlisib (to the dose escalation scheme) plus trastuzumab emtansine 3.6mg/kg IV on day 1 of a 21-day cycle.

DETAILED DESCRIPTION:
This study is a phase Ib open label, single arm, adaptive multi-centre trial. Patients with unresectable locally advanced or metastatic HER2-positive breast cancer who previously received trastuzumab and a taxane, separately or in combination, will be treated with copanlisib plus trastuzumab emtansine 3.6mg/kg IV on day 1 of a 21-day cycle.

3 to 6 patients will be enrolled per dose level. All patients in each level must have completed at least the first cycle of therapy before enrolment in the next dose level begins. Patients not completing the first cycle for a reason other than toxicity will be replaced.

Copanlisib will start at a low level and dose escalations will be performed in cohorts of 3 patients according to a standard 3+3 algorithm.

Dose escalation and determination of maximum tolerated dose (MTD) will be based on occurrences of Dose Limiting Toxicities (DLT).

The first cohort of 3 patients will commence at dose level 1. All patients in each cohort will be observed for one cycle on the specified dose:

* If none of 3 patients at a given dose level experiences a DLT, accrual will continue to the next dose level according to the protocol.
* If 1 of 3 patients experiences a DLT at a given dose level, 3 additional patients will be treated at the same dose. If no additional patient has a DLT in this cohort, accrual will continue to the next dose level according to the protocol.
* If 2 or more patients in 3 or 6 patients treated at a given dose experience a DLT, the dose will be de-escalated to the next lower dose level, which will define the MTD.

If 2 or more patients in 3 or 6 patients treated at the -1 dose level experience DLT, the trial will be stopped.

Primary Objective:

1. To determine the Maximum Tolerated Dose (MTD), for copanlisib in combination with trastuzumab emtansine (T-DM1) in patients with pretreated unresectable locally advanced or metastatic HER2-positive breast cancer.

Secondary Objectives:

1. To evaluate the safety and tolerability of this regimen.
2. To evaluate efficacy measures in patients treated with this regimen.
3. To assess the incidence of cardiotoxicity in patients treated with this regimen.

Exploratory Objectives:

1. To examine for predictive biomarkers in tumour tissue and blood.
2. To examine molecular tumour adaptation to clinical trial therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be provided before any study-specific tests or procedures are performed.
2. Adult women ≥ 18 years of age.
3. Histologically confirmed HER2-positive breast cancer:

   * Documented HER2 overexpression by local laboratory defined as a score of 3+ by IHC or a ratio of ≥ 2.0 by ISH.
   * HER2-positive on diagnostic breast biopsy or surgical breast resection sample or metastatic disease site biopsy.
4. Patient with unresectable locally advanced or metastatic breast cancer who previously received trastuzumab and a taxane, separately or in combination.
5. Patient has received prior therapy for locally advanced or metastatic disease, or developed disease recurrence during or within six months of completing adjuvant therapy.
6. At least one measurable lesion according to RECIST criteria (Version 1.1). Patients with bone only disease are eligible if lesion(s) can be accurately assessed by CT/MRI according to RECIST (Version 1.1).
7. ECOG performance status ≤ 2.
8. Life expectancy of at least 3 months.
9. Availability of fresh tissue and/or archival tumour tissue at screening.
10. Women of childbearing potential must agree to use a highly effective method of contraception when sexually active. This applies from signing of the informed consent form until at least 7 months after the last study drug administration. The investigator or a designated associate is required to advise the patient how to achieve an adequate birth control. Highly effective contraception is defined in the study as methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include:

    i. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).

    ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable and implantable).

    iii. Intrauterine device (IUD). iv. Intrauterine hormone-releasing system (IUS). v. Bilateral tubal occlusion. vi. Successfully vasectomised partner. vii. Sexual abstinence.

    Postmenopausal women defined as follows:
    * Woman 60 years of age or older, OR
    * Woman younger than 60 years of age with spontaneous cessation of menses for at least 12 consecutive months prior to registration, OR
    * Prior bilateral oophorectomy, OR
    * Woman younger than 60 years of age who have had a prior hysterectomy (without bilateral oophorectomy) AND who have an FSH level in the postmenopausal range (or >34.4 IU/L if institutional range is not available).
11. Adequate baseline laboratory values collected no more than 14 days before starting study treatment:

    * Total bilirubin ≤ 1.5 x ULN (< 3 x ULN for patients with metastatic disease in the liver)
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x ULN (≤ 5 x ULN for patients with liver involvement by breast cancer).
    * Lipase ≤ 1.5 x ULN.
    * Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m2 according to the Modification of Diet in Renal Disease (MDRD) abbreviated formula. If not on target, this evaluation may be repeated once after at least 24 hours either according to the MDRD abbreviated formula or by 24 hour sampling. If the later result is within acceptable range, it may be used to fulfil the inclusion criteria instead.
    * International normalized ratio (INR) and partial thromboplastin time (PTT) ≤ 1.5 x ULN. Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior underlying coagulopathy disorder. Close monitoring of these patients (Day 15 of Cycle 1 and Day 1 of each cycle) will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care.
    * Platelet count ≥ 75 x 109/L. For patients with breast cancer bone marrow infiltration, platelet count ≥ 50 x 109/L.
    * Haemoglobin (Hb) ≥ 8 g/dL.
    * Fasting blood glucose ≤6.0 mmol/L if not diabetic or ≤8.9 mmol/L if diabetic.
    * Absolute neutrophil count (ANC) ≥ 1 x 109/L. For patients with malignant bone marrow infiltration, ANC count ≥ 0.75 x 109/L.
12. Left ventricular ejection fraction (LVEF), at or above the Institutions lower limit of normal, as determined by ECHO or MUGA.
13. Patients must have recovered from clinically significant side effects associated with prior radiotherapy and chemotherapy with the exception of fatigue or neuropathy.

Exclusion Criteria:

1. Known breast cancer involvement of the brain, unless adequately controlled based on the clinical judgement of the treating physician.
2. Congestive heart failure > New York Heart Association (NYHA) class II.
3. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before registration.
4. Uncontrolled arterial hypertension despite optimal medical management (per investigator's opinion).
5. Uncontrolled Type I or II diabetes mellitus. Defined as HbA1c > 8.5% as determined during screening laboratory assessments.
6. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before registration.
7. Non-healing wound, ulcer, or bone fracture.
8. Active, clinically serious infections > Grade 2 (CTCAE v5.0).
9. Known history of human immunodeficiency virus (HIV) infection.
10. Hepatitis B (HBV) or hepatitis C (HCV). All patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus laboratory panel Patients who test positive for Hepatitis B surface Antigen (HBsAg) or Hepatitis B core Antigen (HBcAb) will be eligible if they are negative for HBV-DNA; patients who test positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA.
11. Patients with CMV PCR positive.
12. Patients with seizure disorder requiring medication.
13. Patients with evidence or history of bleeding diathesis. Any haemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study treatment.
14. Proteinuria of Grade 3 or higher (CTCAE v5.0). Patient will be excluded if > 2+ on urinalysis (unless 24 hr collection shows 24 hour urinary protein < 3.5g/24hrs).
15. History or concurrent condition of interstitial lung disease of any severity, and/or severely impaired lung functions (as judged by the investigator).
16. Concurrent diagnosis of pheochromocytoma.
17. Pregnant or breast-feeding patients. Women of childbearing potential must have a serum or urine pregnancy test within 7 days of first dose, and a negative result must be documented before start of treatment.
18. Unresolved toxicity higher than CTCAE Grade 1 attributed to any prior therapy/procedure, excluding alopecia, peripheral neuropathy, and bone marrow parameters.
19. Known hypersensitivity to any of the test drugs, test drug classes, or excipients in the formulation.
20. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
21. Any illness or medical conditions that are unstable or could jeopardise the safety of patients and their compliance in the study.
22. Patients permanently withdrawn from study participation will not be allowed to re-enter the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of dose limiting toxicity (DLT) of copanlisib in combination with trastuzumab emtansine within the 1st cycle at each dose level. | 1.5 years

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) is defined as complete response (CR) or partial response (PR) at any time-point on the study; or stable disease (SD) lasting at least 24 weeks based on radiological assessment. | 1.5-2.5 years
Overall Survival (OS). | 1.5-2.5 years
Progression-Free Survival (PFS) assessed according to RECIST criteria version 1.1. | 1.5-2.5 years
Time to Treatment Failure (TTF) is defined as time from registration to discontinuation of therapy or add-on of new anti-cancer therapy for any reason (including death, progression and toxicity). | 1.5-2.5 years
Confirmed tumour response rate as assessed by RECIST criteria version 1.1 | 1.5-2.5 years
Duration of response (DR) as assessed by standard RECIST criteria version 1.1. | 1.5-2.5 years
To evaluate the safety and tolerability of this regimen as measured by incidence of adverse events reported and toxicity evaluation as per the NCI Common Terminology Criteria for Adverse Events (CTCAE version 5.0). | 1.5-2.5 years
To assess the incidence of cardiotoxicity in patients treated with this regimen. | 1.5-2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cancer Trials Ireland Dublin 11, Ireland, Study Director — Cancer Trials Ireland
Locations (3):
- Ireland (2):
  - Cancer Trials Ireland Investigative Site, Cork
  - Cancer Trials Ireland Investigative Site, Dublin
- Cancer Trials Ireland Investigative Site, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided